CLINICAL TRIAL: NCT04349124
Title: Pilot Treatment of Persistent Non-Severe Postpartum Hypertension
Brief Title: Persistent Postpartum Hypertension Pilot Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to continue recruiting
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00104425
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Results first posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Intervention Model Description: Treatment Arm vs Active Control Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Other): The treatment group will be provided with month supply of 30mg tablets of nifedipine extended release prior to discharge from the delivery admission. Dose increases in clinic will be at the discretion of providers, however a treatment algorithm will be provided for guidance.Treatment group will be given a home blood pressure cuff prior to discharge with instructions for use. They will also be scheduled for a 1 week blood pressure check and 4 week postpartum clinic appointment which standard for these patients outside of this proposal.
  Interventions: Drug: Nifedipine Extended-Release Tablets
- Control Group (No Intervention): The control group will not receive any medications at discharge. Providers will be instructed to only prescribe new blood pressure medication at subsequent postpartum visits if the blood pressure is in the severe range (>/=160/110). The control group will be given a home blood pressure cuff prior to discharge with instructions for use. They will also be scheduled for a 1 week blood pressure check and 4 week postpartum clinic appointment which standard for these patients outside of this proposal.

INTERVENTIONS:
Drug: Nifedipine Extended-Release Tablets — Antihypertensive
  Arms: Treatment Group

SUMMARY:
This study is a pilot, open-label, randomized controlled trial of postpartum women with hypertensive disorders pregnancy and persistent non-severe blood pressure. The purpose of the study to provide data that may provide guidance regarding blood pressure management of patients with non-severe postpartum hypertension. There are limited guidelines for best practice with persistent, non-severe hypertension, and treatment in this situation is usually at the provider's discretion.

DETAILED DESCRIPTION:
Study groups will include a treatment with nifedipine extended release or no treatment. Subjects will be randomized 1:1. Subjects randomized to the treatment group will be provided the study drug (nifedipine extended release) at an initial dose of 30mg daily in 1-month supply. The control group will not receive any drug for blood pressure control. the primary outcome is systolic blood pressure at 1 week postpartum.

Subjects in both groups will be scheduled for a 1-week postpartum blood pressure check and routine 4 week postpartum visit. Medication compliance in the treatment group will be assessed via validated questionnaire. The primary outcome of this study is average systolic blood pressure at 1 week postpartum. Patients will be given instructions on blood pressure ranges and specific symptoms when they should contact study staff.

ELIGIBILITY:
Inclusion Criteria:

* Antepartum diagnosis of gestational hypertension
* preeclampsia
* superimposed preeclampsia without antepartum chronic hypertension medication
* Delivery at 23 weeks or greater
* Persistent elevation in BP >24 hours postpartum (>140/90 mm Hg) (2 or more BP >4 hours apart)
* 18 years or older
* English speaking

Exclusion Criteria:

* Need for continuation of antepartum antihypertensive medication
* Contraindication of calcium channel blocker use
* Severe range (160/110 mm Hg) blood pressure requiring treatment >24 hours after delivery
* Requires a 2nd oral antihypertensive medication for blood pressure control inpatient
* Acute cardiomyopathy or heart failure
* Creatinine ≥1.5
* Blood pressure <90/60 within 24 hours of discharge

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenna Hughes, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [29 to 32] | 27 [24 to 32] | 28.5 [26.5 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Average Systolic Blood Pressure at 1 Week Postpartum
Time Frame: 1 week postpartum
Population: Data not collected on 3 participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 4
mmHg | 137.0 (14.5) | 127.3 (7.1)

2. Secondary Outcome: Average Systolic Blood Pressure at 4 Weeks Postpartum
Time Frame: 4 weeks postpartum
Population: Data not collected on 3 participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 4 | 5
mmHg | 130.3 (13.7) | 126.0 (15.6)

3. Secondary Outcome: Average Diastolic Blood Pressure at 1 Week Postpartum
Time Frame: 1 week postpartum
Population: Data not collected on 3 participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 4
mmHg | 89.8 (10.7) | 86.3 (9.2)

4. Secondary Outcome: Average Diastolic Blood Pressure at 4 Weeks Postpartum
Time Frame: 4 weeks postpartum
Population: Data not collected on 3 participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 4 | 5
mmHg | 84.5 (9.8) | 83.2 (10.3)

5. Secondary Outcome: Number of Participants With Blood Pressure < 130/80 mm Hg at 1 Week Postpartum
Time Frame: 1 week postpartum
Population: Data not collected on 3 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 4
Participants
  Yes | 1 | 1
  No | 4 | 3

6. Secondary Outcome: Number of Participants With Blood Pressure < 130/80 mm Hg at 4 Weeks Postpartum
Time Frame: 4 weeks postpartum
Population: Data not collected on 3 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 4 | 5
Participants
  Yes | 1 | 2
  No | 3 | 3

7. Secondary Outcome: Method of Feeding
Time Frame: up to 4 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 5
Participants
  Participants breastfeeding and formula | 2 | 2
  Participants breastfeeding and pumping | 1 | 1
  Participants pumping and formula | 1 | 0
  Participants pumping | 1 | 1
  Participants breastfeeding | 0 | 1

8. Secondary Outcome: Number of Participants With ED/Triage Visits
Time Frame: up to 4 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 5
Participants | 2 | 0

9. Secondary Outcome: Number of Participants With an Increase in Blood Pressure Medication at 1 Week Postpartum
Time Frame: 1 week postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

10. Secondary Outcome: Number of Participants in the no Treatment Group With Initiation of Blood Pressure Medication at 1 Week Postpartum
Time Frame: 1 week postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

11. Secondary Outcome: Number of Participants Who Added a 2nd Blood Pressure Medication at 1 Week Postpartum
Time Frame: 1 week postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Hospital Readmission
Time Frame: up to 4 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 4 weeks postpartum
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT04349124/Prot_SAP_000.pdf